CLINICAL TRIAL: NCT07214194
Title: Vagus Nerve Stimulation to Enhance Memory in Aging
Acronym: VNS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Anthony David Wagner, Professor, Department of Psychology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VNS102025
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Aging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The study will use a sham-controlled, single-blind, within-subject, counterbalanced, randomized design. Each participant will complete four blocks (two active and two sham stimulation) in a counterbalanced within-subject design using an ABBA or BAAB order (A = active taVNS, B = sham stimulation). To ensure equal numbers per order, order will be deterministically assigned by subject ID parity: odd = ABBA, even = BAAB. Subject IDs will be issued sequentially within the age group, yielding balance in both Young and Older groups and effective random assignment of participants to order condition.
Who Masked: Participant
Masking Description: Because the active electrode will be placed on the cymba conchae and the sham on the earlobe, full double-blinding is not feasible; as such, the experimenter will be aware of the active/sham condition status of each experimental block. Participants will be masked/blinded to condition order and hypotheses (they will not be informed which blocks are active vs. sham).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active vagus nerve stimulation (Experimental): Participants will receive active stimulation during memory encoding of picture-word pairs. Active stimulation will occur during two learning phases of the learning and memory task. The total duration of these two phases will be less than 30 minutes.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)
- Sham stimulation (Sham Comparator): Participants will receive sham stimulation during memory encoding of picture-word pairs. Sham stimulation will occur during two learning phases of the learning and memory task. The total duration of these two phases will be less than 30 minutes.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — Non-invasive vagus nerve stimulation will be delivered with a well-validated device. taVNS delivers stimulation on the left ear, with the placement of the stimulating electrode differing between the active and sham conditions. Stimulation will occur during each learning trial (total of 30 trials per phase).

SUMMARY:
The aim of this study is to determine whether non-invasive vagus nerve stimulation enhances memory formation in cognitively healthy older adults and whether the effects of stimulation depend on gut and brain health.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30 years or 65-80 years
* Normal or corrected-to-normal vision (visual acuity)
* Fluent in English

Exclusion Criteria:

* Pregnant
* Symptoms of memory loss
* History of a neurological, psychiatric, or medical condition that could affect cognition or preclude MRI or pupillometry
* Use of medications known to alter cognition
* For older adults, neuropsychological performance that falls outside 1.5 standard deviations of age-adjusted norms and no self-reported memory or attention complaints

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2027-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Recognition Memory (d-prime) | post-active vs post-sham stimulation; up to 2 hours of task
  d' is a signal-detection sensitivity index-how well participants discriminate old (studied) from new (unstudied) items, independent of response bias. Computed as d' = Z(hit rate) - Z(false-alarm rate) from the old/new recognition memory test. Primary analysis is within-person Δhigh-confidence d' (based on "sure old" responses in the 4-point "sure old", "unsure old", "unsure new", "sure new" scale, Δ = active - sham) and Δoverall d' (based on "sure old" and "unsure old" responses). Main comparison is older vs. young, and within the older group also testing moderation by gut-brain axis measures and interactions with preclinical Alzheimer's disease pathology (pTau217, pTau181, Aβ42:40).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Wagner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All other data will be made available via Stanford's Digital Repository (SDR) and will be linked with associated analytic code on the Stanford Memory Lab's Github. Additionally, the task and analysis scripts, along with comments explaining the source code and instructions to install and configure software required to run the scripts, will be shared via the website of the Stanford Memory Lab and our repository on GitHub. SDR is accessible to investigators who are not affiliated with Stanford University and does not require data to be associated with a publication prior to being accepted by the repository. This data archiving approach ensures that the broader scientific community will have long-term access to all data and analysis code.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be made available upon publication of corresponding results or at the end of the award period, whichever is sooner. They will remain available indefinitely or until the end-of-life of the corresponding data-hosting platforms, if no suitable alternative can be identified.
Access Criteria: De-identified MRI and other components of the dataset will be findable and identifiable via persistent Stanford Digital Repository (SDR) URLs. These links will be embedded in published preprints and manuscripts, as well as with direct links on the Stanford Memory Lab's webpage. The SDR does not require data to be associated with a publication to be accepted by the repository. Processed microbiome data tables and metadata will be findable and identifiable through GEO accession numbers. The raw sequencing data will be findable and identifiable through SRA accession numbers.
  Access to de-identified data will not be controlled (i.e., once publicly available, anyone can access the de-identified data).